CLINICAL TRIAL: NCT00926562
Title: A Randomized, Double-blinded Comparison of Iopromide and Iodixanol in Renally Impaired Patients Undergoing Cardiac Catheterization
Brief Title: A Safety Comparison of Iopromide and Iodixanol in Renal Impaired Patients
Acronym: DIRECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Prof. Yundai Chen, Chinese PLA general hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 14147
Record Dates: First submitted 2009-06-19; First posted 2009-06-23 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Kidney Failure, Chronic
Keywords: Contrast Induced Nephropathy; CIN; Cardiac Catheterization
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — iopromide; iodixanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iopromide (Experimental): Drug: Ultravist 370 mgl/ml, injection of intra-artery during cardiac interventional operation
  Interventions: Drug: Iopromide (Ultravist)
- Iodixanol (Active Comparator): Drug: Visipaque 320 mgl/ml, injection of intra-artery
  Interventions: Drug: Iodixanol (Visipaque)

INTERVENTIONS:
Drug: Iopromide (Ultravist) — Iopromide (contrast agent), 370 mgl/ml, an nonionic, monomeric, LOCM
  Other Names: Ultravist
  Arms: Iopromide
Drug: Iodixanol (Visipaque) — Iodixanol (contrast agent) 320 mgl/ml, a nonionic, dimeric, IOCM
  Other Names: Visipaque
  Arms: Iodixanol

SUMMARY:
The investigators intend to find out which contrast agent has less kidney toxicity in renal impaired patients undergoing cardiac angiography or percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
In the diagnosis and treatment of coronary heart disease, patients should undergo cardiac angiography or percutaneous coronary intervention (PCI). In those procedures, the investigators should use the contrast media, and it may cause kidney toxicity especially in the patients with chronic renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Plan to undergo Cardiac Catheterization
* Signed ICF
* eGFR: 30~59 mL/min/1.73m2

Exclusion Criteria:

* Pregnancy
* Under dialysis
* Conditions interfering with Cardiac Catheterization
* Participation in other trials
* Allergic to X-ray contrast media
* Administration of any investigational drug within the previous 30 days
* Intra-arterial or intravenous administration of iodinated contrast medium from 7 days before to 72 hours after the administration of study drug
* Left ventricular ejection fraction (LVEF) less than 30% by ultrasound examination
* Intake of any nephrotoxic medications 24 hours before or after the administration of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients exhibiting a relative increase in serum creatinine >= 50% from baseline. | day 3 postreatment

SECONDARY OUTCOMES:
Proportion of patients developing acute renal failure. | day 30 postreatment
Incidence of a postdose SCr increase ≧25%, a postdose SCr increase ≧1mg/dL, a postdose SCr increase ≧0.5mg/dL, a postdose eGFR decrease ≧25% | days 3

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, MD, Principal Investigator — Chinese PLA General Hospital
Locations (19):
- China (19):
  - Beijing CHAO-YANG Hospital, Beijing, Beijing Municipality
  - General Hospital of Armed Police Forces, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Shi Jing Shan Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Chinese PLA general hospital, Beijing, Beijing Municipality
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - The Second Hospital of Xiangya, Changsha, Hunan
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jinlin
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Renji Hospital affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Changhai Hospital affiliated to the second millitary medical university, Shanghai, Shanghai Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Teda International Cardiovascular Hospital, Tianjin, Tianjin Municipality
  - The Second Hospital Affiliated to Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital affiliated to Zhejiang, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Chen Y, Hu S, Liu Y, Zhao R, Wang L, Fu G, He Q, Su X, Zheng Y, Qi X, Liu H, Wang J, Gao W, Wang M, Liu S, Zheng X, He B, Yang P, Zhou S, Gao C, Qiu C. Renal tolerability of iopromide and iodixanol in 562 renally impaired patients undergoing cardiac catheterisation: the DIRECT study. EuroIntervention. 2012 Nov 22;8(7):830-8. doi: 10.4244/EIJV8I7A126. PMID 23045301